CLINICAL TRIAL: NCT06261255
Title: Efficacy of Digitally Tooth Autotransplantation With Adjunctive Use of Enamel Matrix Derivatives (EMD): A Prospective Case Series
Brief Title: Autotransplantation and Enamel Matrix Derivatives Case Series
Acronym: ATTCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Ignacio Pedrinaci Peñalver, Dr. Principal investigator, Universidad Complutense de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATT_CS
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Tooth Loss
Keywords: emdogain; enamel matrix derivatives; tooth autotransplantation; tooth autogenous transplantation; digital planning
MeSH Terms: conditions — Tooth Loss | interventions — emerin

STUDY DESIGN:
Intervention Model Description: This clinical investigation is a single-center, prospective case series study and is reported in compliance with the Preferred Reporting of Case Series in Surgery (PROCESS) guidelines. The study was conducted at the Department of Periodontology of the University Complutense of Madrid between March 2021 and September 2023.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATT + EMD (Experimental): There is only 1 arm, autotransplantation (ATT) + adjunctive EMD
  Interventions: Procedure: ATT + EMD

INTERVENTIONS:
Procedure: ATT + EMD — All surgical treatments will be performed by the same experienced periodontist (IP) after the administration of local anesthesia. Initially, tooth sectioning of the hopeless tooth (receptor) will be carried out using fissure carbide burs, and the remaining fragments will be extracted as minimally invasively as possible. A tooth-supported surgical guide will be used to prepare the recipient site following the 3D planning. Additional alveoloplasty procedures will be performed with round diamond burs if necessary to adapt the CARP model to the virtual planning position. The donor tooth will be extracted as atraumatically as possible, utilizing a piezoelectric surgical instrument if osteotomy is required, and avoiding the use of elevators or forceps over the root surface. Extraorally, EMD will be applied to the root surface of the donor tooth

SUMMARY:
The goal of this prospective case series is to compare the adjunctive use of enamel matrix derivatives in the treatment of tooth autotransplantation in terms of clinical attachment level.

The main question it aims to answer is:

- What is the benefit, in terms of clinical attachment level, of using enamel matrix derivatives adjunctive to tooth autotransplantation?

Participants will be subjected to a digitally protocol of tooth autotransplantation.Only one group (test) is assessed. It will be supplemented with the application of enamel matrix derivatives before the placement of the transplanted tooth into the surgically produced alveolus.

DETAILED DESCRIPTION:
All surgical treatments will be performed by the same experienced periodontist (IP) after the administration of local anesthesia. Initially, tooth sectioning of the hopeless tooth (receptor) will be carried out using fissure carbide burs, and the remaining fragments will be extracted as minimally invasively as possible. A tooth-supported surgical guide will be used to prepare the recipient site following the 3D planning. Additional alveoloplasty procedures will be performed with round diamond burs if necessary to adapt the computed aid rapid prototyping (CARP) model to the virtual planning position. The donor tooth will be extracted as atraumatically as possible, utilizing a piezoelectric surgical instrument if osteotomy is required, and avoiding the use of elevators or forceps over the root surface. Extraorally, EMD will be applied to the root surface of the donor tooth.

After positioning the donor tooth onto the surgically created recipient bed, a semi-rigid orthodontic wire will be used to splint the tooth to the mesial and distal adjacent teeth, and sutures will be applied to closely adapt the soft tissues around the autotransplanted tooth. Occlusal adjustments will be made if necessary. Alternatively, orthodontic composite bite stops will be placed on top of adjacent teeth to obtain temporary dental disocclusion.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years old) capable of providing informed consent, teeth deemed unrestorable and in need of replacement
* presence of a viable, healthy, periodontally stable, and nonfunctional tooth (e.g., third molar) suitable for autotransplantation
* periodontally healthy individuals or those with stable periodontal conditions after periodontal therapy.

Exclusion Criteria:

* clinical attachment loss of the donor teeth
* compromised general health or patients with systemic diseases that could influence the therapy outcome (uncontrolled diabetes mellitus, bone disorders, etc.)
* pregnant or nursing women
* chronic use of corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or immune-modulator drugs
* patients requiring medications that affect bone metabolism (bisphosphonates)
* chronic oral mucosa diseases
* evident signs of severe bruxism or clenching habits
* smokers of more than 10 cigarettes per day
* non-compliant patients with 25% plaque index at the time of re-evaluation after non-surgical periodontal therapy and oral hygiene instructions
* patients unable to attend study-related procedures and follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | through study completion, an average of 1 year
  CAL level changes on the donor tooth between the baseline situation and the last follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Pedrinaci, DDS, Principal Investigator — Universidad Complutense de Madrid
Locations (2):
- Spain (2):
  - Universidad Complutense de Madrid, Madrid
  - Universidad Complutense Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No